CLINICAL TRIAL: NCT02391701
Title: Effect of an Atlantic Diet on Anthropometric Indices and Serum Lipid Profile in a General Population: a Randomised Controlled Trial
Brief Title: Effect of an Atlantic Diet on Anthropometric Indices and Serum Lipid Profile
Acronym: GALIAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Maria del Mar Calvo Malvar, Pharmacy PhD, Specialist in Laboratory Medicine, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCSantiago
Record Dates: First submitted 2015-02-11; First posted 2015-03-18 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Disease; Adiposity; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Hypercholesterolemia | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet group (Experimental): Diet program 1 day a month for 3 months in 120-minute diet sessions + Freely they receive AD food: vegetables, cheese, olive oil, mussels and wine.
  Interventions: Behavioral: Diet
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Diet — diet program 1 day a month for 3 months in 120-minute diet sessions + freely receive Atlantic Diet food (vegetables, cheese, olive oil, mussels and wine)
  Arms: Diet group

SUMMARY:
BACKGROUND:

The Southern European Atlantic Diet (SEAD) is the traditional diet of Northern Portugal and Galicia, a region in northwest Spain. The SEAD has been associated with a lower risk of non-fatal acute myocardial infarction. Possible mechanisms of this association may be related with a lower concentration of markers of inflammation and with reduced triglycerides, insulin, insulin resistance, and systolic blood pressure.

Aim: To evaluate the effect of an Atlantic Diet on i) lipid profile, ii) markers of inflammation, and iii) anthropometric indices in a population-based study

METHODS:

This is a non-pharmacological clinical trial study which is performed on a family-oriented basis. 250 families (~ 750 children and adults, older than 3 years) were selected to participate in the study and randomized into Atlantic Diet (AD) (n=125 families) and control (n=125 families) groups. The AD groups participate in a diet program 1 day a month for 3 months in 120-minute diet sessions and freely receive AD food, characterized by a high intake of vegetables, cheese, olive oil, mussels and by wine consumption during meals. Control group subjects do not participate in any regular diet activity during this period and did not receive additional food. Exclusion criteria are alcoholism, lipid treatment, dementia, and terminal disease.

Weight, BMI, waist circumference (WC), skin folds, nutrient intake from 3-day recalls, food frequency questionnaire, physical activity, blood pressure, metabolic function (fasting blood glucose, HBA1c, insulin resistance and lipid profile), and inflammation markers (c-reactive protein, interleukin 6 and tumor necrosis factor-alpha) are measured at baseline, 3 and 6 months. Mixed effect models will be performed to assess the significance of changes in the cardiometabolic parameters.

The primary end point is the change in lipid profile compared with baseline and the control group arm at the end of Month 6. The secondary exploratory end points were change in anthropometric indices and inflammation markers at Month 6.

DETAILED DESCRIPTION:
The intervention period lasted 6 months. At the baseline visit all AD subjects received information on the Atlantic diet and how to follow it; the nutritionists' messages were adapted to the clinical condition of each subject, his/her preferences, needs, beliefs and culture. Special care was taken with patients who were obese, had diabetes or who had high blood cholesterol; conflicts with recommendations made by subjects' own doctors or nutritionists were avoided. All questionnaires (see below) were filled out in the presence of the nutritionists, except for 3-day food records which the subjects handed in completed. The latter were reviewed in the presence of the subjects in order to correct any errors or add missing information. At the 3 and 6 month visits, the nutritionists reminded the subjects about the Atlantic diet and the helped them complete their questionnaires.

Foods were provided to the families of the AD group. Wine was provided only to non-tee-total adults. Food packages were delivered every three weeks to the family home. The food included in the package was calculated for the total number of family members, even if not all were taking part in the study. At delivery, a form was filled in to verify that the previous lot of food had been consumed, and to note any problems.

ELIGIBILITY:
A random sample of the population 18 years and older was drawn from the National Health System Register in order to select the index subjects.These individuals (index subjects) and all family members sharing the same house were invited to participate in the study.

Inclusion Criteria:

1. For the index subject:

   * Female or male.
   * 18 years and older.
   * Living in a family unit with two or more people.
2. For the other family members:

   * Female or male.
   * Age between 3 to 85 years.

Exclusion Criteria:

1. For the index subject:

   * Alcoholism
   * Lipid treatment
   * Pregnant
   * Major cardiovascular disease
   * Dementia
   * Terminal disease
2. For the other family members:

   * Alcoholism
   * Pregnant
   * Major cardiovascular disease
   * Dementia
   * Terminal disease

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mar Calvo, PhD, Study Chair — Servicio Galego de Saude (SERGAS)
Locations (1):
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cambeses-Franco C, Gude F, Benitez-Estevez AJ, Gonzalez-Garcia S, Leis R, Sanchez-Castro J, Moreira MT, Feijoo G, Calvo-Malvar M. Traditional Atlantic Diet and Its Effect on Health and the Environment: A Secondary Analysis of the GALIAT Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2354473. doi: 10.1001/jamanetworkopen.2023.54473. PMID 38324314
- [Derived] Calvo-Malvar Mdel M, Leis R, Benitez-Estevez AJ, Sanchez-Castro J, Gude F. A randomised, family-focused dietary intervention to evaluate the Atlantic diet: the GALIAT study protocol. BMC Public Health. 2016 Aug 18;16(1):820. doi: 10.1186/s12889-016-3441-y. PMID 27539113

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diet Group | Control
Started | 367 | 353
Completed | 346 | 315
Not Completed | 21 | 38

BASELINE CHARACTERISTICS:
Population: Data updated from the review of the data collection notebooks.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Group | Control | Total
Number analyzed (Participants) | 367 | 353 | 720
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80 | 66 | 146
  Between 18 and 65 years | 238 | 255 | 493
  >=65 years | 49 | 32 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (19.8) | 40.2 (20.8) | 39.4 (20.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 211 | 425
  Male | 153 | 142 | 295
Region of Enrollment [Number; unit: participants]
  Spain | 367 | 353 | 720

OUTCOME MEASURES:

1. Primary Outcome: Changes in Total-cholesterol Levels
Description: Change from baseline in total cholesterol:
  Enzymatic method using standard kits on an Advia 2400 Clinical Chemistry System (Siemens Healthcare Diagnostics) [Time Frame: 6 months ]
Time Frame: baseline and 6 months
Population: Intent to treat population (all participants who were randomized)
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Diet Group | Control
Number analyzed (Participants) | 367 | 353
mg/dl | -6.9 [-9.3 to -4.5] | -0.6 [-3.1 to 2.0]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Measurements will be made in triplicate and recorded by standard methods using a SECA 813 digital balance with the subjects in underwear and barefoot. Body weight will be measured to the nearest 0.1 kg.
Time Frame: Baseline and 6 months
Population: Intent to treat population (all participants who were randomized)
Measure: Mean (95% Confidence Interval); unit: Kg
Arm/Group | Diet Group | Control
Number analyzed (Participants) | 367 | 353
Kg | -0.32 [-0.62 to -0.01] | 0.62 [0.33 to 0.91]

3. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: BMI will be calculated as body weight (kg) divided by height (m) squared. The BMI of subjects under 18 years of age will be standardised using World Health Organization (WHO) reference data.
Time Frame: Baseline and 6 months
Population: Intent to treat population (all adult participants who were randomized). The BMI of subjects under 18 years of age were not included (80 participants in the Diet Group and 66 participants in the Control Group).
Measure: Mean (95% Confidence Interval); unit: Kg/m2
Arm/Group | Diet Group | Control
Number analyzed (Participants) | 287 | 287
Kg/m2 | -0.29 [-0.43 to -0.16] | 0.17 [0.04 to 0.29]

4. Secondary Outcome: Change From Baseline in Hip/Waist Index
Description: Waist circumference will be measured at the narrowest point between the bottom rib and the top of the iliac crest using a SECA 201 flexible, non-elastic tape.
  Hip circumference will be measured at the point of greatest prominence of the gluteal muscles using a SECA 201 flexible, non-elastic tape.
Time Frame: Baseline and 6 months
Population: Intent to treat population (all participants who were randomized)
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Diet Group | Control
Number analyzed (Participants) | 367 | 353
Ratio | -0.015 [-0.020 to -0.010] | -0.003 [-0.008 to 0.001]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Enzymatic method using standard kits on an Advia 2400 Clinical Chemistry System (Siemens Healthcare Diagnostics)
Time Frame: Baseline and 6 months
Population: Intent to treat population (all participants who were randomized)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Diet Group | Control
Number analyzed (Participants) | 367 | 353
mg/dL | -1.9 [-2.9 to -0.9] | -2.6 [-3.6 to -1.6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Diet Group | Control
All-Cause Mortality (participants affected / at risk) | 0/367 | 0/353
Serious Adverse Events (participants affected / at risk) | 0/367 | 0/353
Other Adverse Events (participants affected / at risk) | 0/367 | 0/353

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No